CLINICAL TRIAL: NCT00639951
Title: Multicentric, Randomized,Controlled and Comparative Study to Evaluate the Efficacy of Two Treatment Schemes With Antivipmyn ® for the Treatment of Snake Bite Envenomation
Brief Title: Study to Evaluate the Efficacy of Two Treatment Schemes With Antivipmyn ® for the Treatment of Snake Bite Envenomation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Administrative reasons
Sponsor: Instituto Bioclon S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YA-07/01
Record Dates: First submitted 2008-03-13; First posted 2008-03-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Snake Bite
Keywords: Snake Bite; Antivenin Treatment
MeSH Terms: conditions — Snake Bites | interventions — antivipmyn Africa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A Normal dose Group (Active Comparator): 20 vials up front in a Single Dose of Antivipmyn in 500 ml of solution IV, administered in 60 minutes. After 12 hours, it has to be perfomed a clinical evaluation of the patient. Each patient is going to have clinical studies of coagulation time and also the fibrinogen measures, this at 2, 4, 6, 8, 10, 12, 48, 72, 96 hours.All patients who have received at least one dose of medication study will be contacted by telephone to investigate the presence of symptoms suggestive of continuing with effect snake venom, or the presence of an adverse event, or any signs or symptoms indicating the presence of a hypersensitivity response to Antivipmyn® including serum sickness. If symptoms suggestive of an adverse event were discovered, the patient will referred for appropriate treatment.
  Interventions: Biological: A
- B Placebo Group (Placebo Comparator): 20 vials fractionated into 4 doses of 5 vials each of Antivipmyn ®. The treatment schedule for each subject is a dose of 5 vials Antivipmyn® every 2 hours to complete 20 vials, the total duration is 6 hours of the treatment. Each dose IV shall apply in physiological solution 250ml, and finish its application in 15 minutes. For pediatric patients the volume administered should not exceed the recommended fluid volume according to your body weight. After the assessment at 12 hours, it can be administered at the discretion of more antivenom attending by the physician.
  Interventions: Biological: Antivipmyn ®

INTERVENTIONS:
Biological: A — 20 vials up front in a Single Dose of Antivipmyn
  Other Names: Crotalinae (pit viper) equine immune F(ab)2
  Arms: A Normal dose Group
Biological: Antivipmyn ® — 20 vials fractionated into 4 doses of 5 vials each of Antivipmyn ®
  Other Names: Crotalinae (pit viper) equine immune F(ab)2
  Arms: B Placebo Group

SUMMARY:
The purpose of this study is to compare whether a same total dose given up front as a single dose is more effective and as safe as the same dose given as a fractioned dose.

Evaluate the Utility of the the Dry Tube Test Evaluating its Correlation with Coagulation Test Results (fibrinogen, platelets, INR, PT and PTT).

Explore the Evolution of some Serum Markers (CK, DHL, metalloproteinase), Amount of Venom and Antivenom Levels and the Progression of Local Lesions.

DETAILED DESCRIPTION:
Snake bite Envenomation is a Public Health Problem especially for tropical and subtropical countries. The WHO estimates 40 000 annual deaths in the world for this cause. In México the Ministry of Health estimated 3 882 cases on 2005, being the age of 15-44 the most affected. There are not official numbers of mortality, although the thought is that there are few cases of death, most of them related with a delay on treatment.

There are a broad variety of clinical presentations depending on many factors such as species, snake bite variability or patient conditions. Proteolytic action of venom produces amines and vasoactive peptides such as bradykinin, histamine and serotonin which cause capillary lesions with anticoagulant effects. Coagulopathy is one of the most important systemic consequences. The Dry Tube Test has been proposed as an indirect test to evaluate coagulopathy related to this pathology.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 6 to 65 years of age
* Presenting for emergency treatment of snake bite
* Requiring treatment with antivenom
* Informed consent document read and signed by patient (or parent/legal guardian)
* Participation within the last month on any clinical trial
* Arrival to Hospital within 24 hours after the snake bite

Exclusion Criteria:

* Allergy to horse serum
* Underlying medical conditions that significantly alter coagulation (oral anticoagulants, vitamin K deficiency, hepatic disease)
* Use of AINE 48 hours previously
* Use of any antivenom 2 weeks previously
* Pregnancy or breast-feeding women

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Resolution of systemic signs and symptoms of snake bite envenomation expressed as % of patients requiring additional antivenom and % of patients that are stable | 12 hours after initial treatment

SECONDARY OUTCOMES:
Evaluate the correlation between Dry Tube Test and Coagulation Test (PT, INR, PTT, platelets and fibrinogen) | baseline, 2,4,6 hours and after each extra dose of Antivenom
Evaluate Venom and Antivenom Levels with the other parameters | baseline, 2 hours after initial treatment and after each extra dose of Antivenom
Evaluate the possible relation of the serum markers (LDH, CPK, metalloproteinases)and local damage evolution. | baseline, 2, 4,6 and after each extra dose of Antivenom

CONTACTS AND LOCATIONS:
Overall Officials: Walter García, MD, Study Director — Instituto Bioclon; Anabel Loza, MD, Study Chair — Instituto Bioclon
Locations (5):
- Mexico (5):
  - Hermosillo Site, Sonora, Hermosillo
  - Nayarit Site, Tepic, Nayarit
  - Hospital Universitario de la UANL "Dr. José Eleuterio González", Monterrey, Nuevo León
  - Ciudad Valles Site, Ciudad Valles, San Luis Potosí
  - Tempoal Site, Tempoal de Sánchez, Veracruz

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided